CLINICAL TRIAL: NCT02612181
Title: The Effect of Dexmedetomidine on Microcirculation in Septic Shock- A Double-blinded Study
Brief Title: Dex on Microcirculation in SS-A Double-blinded Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, Principal investigator, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015ZDSYLL016.1
Record Dates: First submitted 2015-11-17; First posted 2015-11-23 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Septic Shock
Keywords: dexmedetomidine; microcirculation; septic shock
MeSH Terms: conditions — Shock, Septic | interventions — Dexmedetomidine; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine group (Experimental): Dexmedetomidine group: Dexmedetomidine infusion for dexmedetomidine group to the goal of sedation: Richmond agitation-sedation scale 0 to -2 Dexmedetomidine doses 0-0.7 mcg/kg/h
  Interventions: Drug: Dexmedetomidine for dexmedetomidine group
- Control group (Placebo Comparator): Control group: Placebo infusion for control group to the goal of sedation: Richmond agitation-sedation scale 0 to -2 Control drug doses 0-0.7 mcg/kg/h
  Interventions: Drug: Dexmedetomidine for dexmedetomidine group

INTERVENTIONS:
Drug: Dexmedetomidine for dexmedetomidine group — The effect of dex and placebo for sedation on microcirculation
  Other Names: Placebo for control group

SUMMARY:
The investigators preliminary study showed that dexmedetomidine might improve microcirculation in septic shock patients. To test this effect, the investigators will conduct double-blinded study.

DETAILED DESCRIPTION:
Dexmedetomidine is a highly selective α2-adrenoreceptor agonist for sedation of adult critically ill patients which exhibits sedative and analgesic effects. Recent studies suggest that dexmedetomidine to restore adrenergic vasoconstrictor responsiveness in septic shock, and prevents alterations of pain rat model intestinal microcirculation Induced by surgical stress，even it can reduce the mortality of endotoxemic rats and patients with severe sepsis. The investigators preliminary study showed that dexmedetomidine might improve microcirculation in septic shock patients. To test this effect, the investigators will conduct double-blinded study.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock patients despite early goal directed therapy
* Agree to participate this study

Exclusion Criteria:

* Age< 18
* Pregnancy
* Bradycardia (HR<55bpm)
* Systolic Blood Pressure < 80 mmHg / Mean arterial pressure < 50 mmHg on maximal support
* Death imminent
* Unlikely to survive 90 days
* Acute liver failure
* Dementia
* High-grade block in the absence of a functioning pacemaker.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Microcirculatory function as assessed by Microvascular flow index | 30 minutes
  sedation for 30 minutes then monitor the microcirculation

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided